CLINICAL TRIAL: NCT01087307
Title: Sample Collection Registry for Quality Control of Biological and Environmental Specimens and Assay Development and Testing
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100063; 10-E-0063
Record Dates: First submitted 2010-03-13; First posted 2010-03-16 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12-15

CONDITIONS: Exposure
Keywords: Serum; Urine Collection; Saliva; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adult Volunteer: Healthy adult volunteer

SUMMARY:
Background:

- Researchers are interested in developing a registry protocol to obtain biologic and environmental samples anonymously from adult volunteers for use in laboratory tests and studies. The samples will be used to determine if new tests are sufficiently valid and precise to be used in research studies and for quality control purposes.

Objectives:

- To provide a registry of samples for test development, validation, analysis, and quality control at the National Institute of Environmental Health Sciences.

Eligibility:

- Male and nonpregnant female volunteers at least 18 years of age.

Design:

* Samples to be collected will include blood, urine, saliva, household dust, cheek cells, hair, nasal cells, stool, nail clippings, exhaled breath condensate, or sperm.
* Specimens may be collected during a one-time sample collection, or participants may be asked to provide specimens on several occasions over a specified period, not to exceed 1 year.
* Eligible participants will be asked to come to the clinical research unit to have their blood drawn and any noninvasive samples retrieved. Prior to blood draw, researchers will administer a brief past 24-hour questionnaire for research purposes. Specimens will be collected using standard clinical protocols.
* Participants will receive monetary compensation for providing samples for this protocol.

DETAILED DESCRIPTION:
We propose a sample collection registry protocol for use in obtaining biologic and environmental samples anonymously from adult volunteers for use in laboratory assay evaluation. The samples will be used to determine if new tests are sufficiently valid and precise to be used in research studies and for quality control purposes. In studies involving the storage and analysis of laboratory specimens, it is essential to evaluate the performance of available assays and to actively assess the impact of storage and handling on the quality of samples and laboratory analyses. Specifically, it is essential to 1) demonstrate that an assay is sufficiently reproducible and stable over time such that differences in levels among individuals in the population can be detected; 2) evaluate assay reliability by sending blinded anonymous samples along with study samples to testing labs for quality control purposes; 3) test proposed laboratories or methods by using replicate samples from the population in order to choose the laboratory or method with the greater precision, and; 4) assess how sample collection, handling, and storage procedures affect measured levels of specific analytes to allow for informed decisions about whether to proceed with a specific analysis. Under this protocol, assays could include evaluation of immunologic parameters, genes and gene products, peptides, proteins, hormones, lipids, viability of cells, evaporation and dilution effects, chemical toxins and their metabolites, micronutrients, metals and more. For some samples, lymphocytes will be extracted for use in studies of lymphocytes and/or immortalized cells. Samples to be collected will include blood, urine, saliva, household dust, cheek cells, hair, nasal cells, stool, nail clippings, exhaled breath condensate, sperm samples, skin cells, and/or sputum. In addition, a pulmonary function test (PFT) may be conducted to collect lung function information. Since it is important to collect samples from the general population, this protocol covers collection of samples from non-pregnant adults (male and female, age 18+). Specimens may be collected during a one-time sample collection, or participants may be asked to provide specimens on several occasions over a specified period, not to exceed one year.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

All participants must be non-pregnant and 18 years of age or older. No children, cognitively impaired persons, or prisoners will be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 5326 (Actual)
Dates: Start 2010-03-02 (Actual)

PRIMARY OUTCOMES:
The endpoint is to create a biobank of samples which can be used for development and optimization of assays. | 24 hours
  The objective of each collection is to generate a small pool of biological or environmental samples with which to develop and test specific laboratory assays, to maintain freezer and specimen handling quality control, to have blinded quality control specimens for testing labs, and to assess exposure variability over time.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Kirschner, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to make IDP available to others.

REFERENCES:
- [Derived] Whitehead GS, Hussain S, Fannin R, Trempus CS, Innes CL, Schurman SH, Cook DN, Garantziotis S. TLR5 Activation Exacerbates Airway Inflammation in Asthma. Lung. 2020 Apr;198(2):289-298. doi: 10.1007/s00408-020-00337-2. Epub 2020 Feb 14. PMID 32060608
- [Derived] Hussain S, Johnson CG, Sciurba J, Meng X, Stober VP, Liu C, Cyphert-Daly JM, Bulek K, Qian W, Solis A, Sakamachi Y, Trempus CS, Aloor JJ, Gowdy KM, Foster WM, Hollingsworth JW, Tighe RM, Li X, Fessler MB, Garantziotis S. TLR5 participates in the TLR4 receptor complex and promotes MyD88-dependent signaling in environmental lung injury. Elife. 2020 Jan 28;9:e50458. doi: 10.7554/eLife.50458. PMID 31989925
- [Derived] Saini N, Roberts SA, Klimczak LJ, Chan K, Grimm SA, Dai S, Fargo DC, Boyer JC, Kaufmann WK, Taylor JA, Lee E, Cortes-Ciriano I, Park PJ, Schurman SH, Malc EP, Mieczkowski PA, Gordenin DA. The Impact of Environmental and Endogenous Damage on Somatic Mutation Load in Human Skin Fibroblasts. PLoS Genet. 2016 Oct 27;12(10):e1006385. doi: 10.1371/journal.pgen.1006385. eCollection 2016 Oct. PMID 27788131
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-E-0063.html